CLINICAL TRIAL: NCT00003576
Title: Surgery and Adjuvant Radiotherapy Versus Concurrent Chemo-Radiotherapy for Resectable (Non-Metastatic) Stage III/IV Head and Neck Squamous Cell Cancer
Brief Title: Surgery and Radiation Therapy Compared With Chemotherapy and Radiation Therapy in Treating Patients With Stage III or Stage IV Head and Neck Cancer That Can Be Removed During Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066643; NMRC-SHN01; EU-97015
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2007-04

CONDITIONS: Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin; Fluorouracil; Surgical Procedures, Operative; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: fluorouracil
Procedure: surgical procedure
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known whether surgery plus radiation therapy is more effective than chemotherapy plus radiation therapy for head and neck cancer.

PURPOSE: This randomized phase III trial is studying surgery and radiation therapy to see how well they work compared to chemotherapy and radiation therapy in treating patients with stage III or stage IV head and neck cancer that can be removed during surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the complete response rate, disease-free survival, and overall survival of patients with resectable (nonmetastatic) stage III or IV squamous cell cancer of the head and neck treated with surgery and adjuvant radiotherapy versus concurrent chemo-radiotherapy.

OUTLINE: This is a randomized study. Patients are stratified according to primary site of disease (oral cavity/oropharynx vs larynx/hypopharynx vs others) and nodal status (node negative vs positive).

* Arm I: Patients undergo resection of the tumor, followed no more than 6 weeks later by radiotherapy to the primary tumor and upper neck once a day, 5 days a week, for 6 weeks.
* Arm II: Patients undergo radiotherapy in addition to chemotherapy with fluorouracil and cisplatin. Radiotherapy is given once a day, 5 days a week, for 6.5 weeks to the primary tumor and upper neck. Fluorouracil and cisplatin are administered by continuous infusion for 4 days beginning on day 1 of the first week of radiotherapy. A second course of fluorouracil and cisplatin is given on day 28.

Patients who have failed or are suspected to have failed chemo-radiotherapy should be considered for salvage surgery.

Patients are followed once a month for the first year, every 2 months for the second year, every 3 months for the third year, and every 6 months thereafter.

PROJECTED ACCRUAL: Approximately 200 patients will be accrued over a 4-5 year period.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed head and neck squamous cell cancer (excluding nasopharynx and salivary glands) on biopsy of the primary lesion or the neck mass
* Stage III or IV disease

  * No evidence of distant or systemic metastases
* Resectable disease

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* WBC greater than 3000/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* SGOT less than 2 times upper limit of normal
* Bilirubin less than 1.4 mg/dL

Renal:

* Creatinine less than 1.6 mg/dL

Other:

* No prior or concurrent primary malignancies
* Not pregnant
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy to the head and neck

Surgery:

* See Disease Characteristics
* No prior surgery (other than biopsy)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 1997-01; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Response at 6 weeks after completion of study treatment
Disease-free survival
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Soo Khee Chee, MD, Study Chair — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre - Singapore, Singapore, Singapore

REFERENCES:
- [Result] Soo KC, Tan EH, Wee J, Lim D, Tai BC, Khoo ML, Goh C, Leong SS, Tan T, Fong KW, Lu P, See A, Machin D. Surgery and adjuvant radiotherapy vs concurrent chemoradiotherapy in stage III/IV nonmetastatic squamous cell head and neck cancer: a randomised comparison. Br J Cancer. 2005 Aug 8;93(3):279-86. doi: 10.1038/sj.bjc.6602696. PMID 16012523